## **CONSENT FORM**

## 1/9/14

for

Group-based Intervention for Club Patrons (AA022331, NCT03652688)

Principal Investigator:

Brenda A. Miller, Ph.D., Prevention Research Center, PIRE, Berkeley, CA

Co-Investigators:

Hilary Byrnes, Ph.D., Prevention Research Center, PIRE, Berkeley, CA
Beth Bourdeau, Ph.D., Prevention Research Center, PIRE, Berkeley, CA
Joel Grube, Ph.D., Prevention Research Center, PIRE, Berkeley, CA
David Buller, Ph. D., Klein Buendel, Golden, CO.

## **Project Coordinator:**

Veronica Rogers, B.S., Prevention Research Center, PIRE, Berkeley, CA

## **Consent Form**

We are from the Pacific Institute for Research and Evaluation and we are conducting interviews to learn more about how we can improve safety at dance events such as the one you are attending tonight. We need information from people like you to do this. We are **not** associated with any law enforcement agency and we are **not** associated with any media organization. The organizers know we are here and have given their permission for us to be here but we are not working for the organizers or otherwise affiliated with the organizers, owners, or venue operators. You were selected completely by chance and you are being asked to **VOLUNTARILY PARTICIPATE** in this study.

WE WILL NOT ASK FOR YOUR NAME AND ALL OF YOUR INFORMATION IS ANONYMOUS. We will ask you a few questions about yourself (e.g., age, residential zip code), your prior attendance at dance events, your experiences at tonight's events, including some questions on sexual experiences, and your use of tobacco, alcohol, over-the-counter drugs, and other drugs. We will collect a sample of your saliva and your breath for later analysis. We will NOT know the results of this analysis tonight. THE RESULTS CAN IN NO WAY BE ASSOCIATED WITH YOU. There is a possibility that some question or questions may make you uncomfortable. You do have the right to refuse to answer any question and the right to withdraw from the study at any time. No one will be able to connect your survey responses or your results from the saliva or breath test with you because this information is collected anonymously.

Based upon the information that we obtain from this study, our goal is to work with the organizers and owners to improve safety for people attending future dance events.

We will give you \$15 for your participation--\$ 5 on your way into the event and \$10 on your way out.

You may ask the interviewers any questions about the study you may have. You may also contact the Principal Investigator, Dr. Brenda A. Miller, Prevention Research Center/PIRE, 1995 University Avenue, Suite 450, Berkeley, CA 94704; telephone 510 883-5768; email: <a href="mailto:bmiller@prev.org">bmiller@prev.org</a> or Co-Principal Investigator, Dr. Debra Furr-Holden, PIRE, 11720 Beltsville Dr., Suite 900, Calverton, Md. 20705; telephone 310 755-2718; email: <a href="mailto:dfurr-holden@pire.org">dfurr-holden@pire.org</a>. If you have questions about your rights as a participant in a research study, you may contact Elysia Oudemans, Manager of Research Integrity Compliance, Pacific Institute for Research and Evaluation, 11720 Beltsville Drive, Suite 900, Calverton, MD 20705; toll free 1-866-PIRE-ORG, ext 2757; email: oudemans@pire.org. This study is funded by the National Institutes of Health.

Thanks for your time!

Group-based Intervention for Alcohol, Drugs and Aggression among Club Patrons, B.A. Miller, PI, Group based consent form\_RCT Sample, 1/9/14